CLINICAL TRIAL: NCT06624735
Title: Behavioral Changes Among Asthmatic Children in Sohag Universty Hospital
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Aya Ezeldin Abdelmotgaly, Resident-pediatric department-sohag hospital university, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: soh-Med-24-07-04MS
Record Dates: First submitted 2024-08-28; First posted 2024-10-03 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Bronchial Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cases group (Active Comparator): Children aged 4-12 years Confirmed diagnosed as asthma
  Interventions: Diagnostic Test: psychometry
- control group (Active Comparator): Children below age of 4 years and aboveage of 12 years . not Diagnosed with any other chronic medical conditions
  Interventions: Diagnostic Test: psychometry

INTERVENTIONS:
Diagnostic Test: psychometry — ADHD test and measurement of IQ level

SUMMARY:
Asthma is considered the most common chronic childhood disease and mainly affects children resident in urban areas. Asthma has been designated a serious public health problem due to the increase in its prevalence over the last two decades and the associated high health service costs in admissions and hospitalizations The cause of asthma is not yet completely understood, and there is no consensus about its etiology. A vast body of research emphasizes the role of genetic and environmental factors in the appearance of asthma, and a great deal of interest has recently emerged concerning the relationship between psychosocial factors and asthma morbidity Behavioural problems in children are generally described as "internalizing", which includes "anxiety, depressive, and somatic symptoms" or "externalizing", which includes "oppositional, hyperactive conduct". Both internalizing and externalizing problems can be experienced by healthy children with abnormal and "borderline" personality disorder, the latter referring to a mental illness marked by an ongoing pattern of varying moods, self-image, and behaviour

ELIGIBILITY:
Inclusion Criteria:

Children aged 4-12 years Confirmed diagnosed as asthma

Exclusion Criteria:

Children below age of 4 years and aboveage of 12 years . Diagnosed with any other chronic medical conditions (e.g., cardiac , liver , renal and other chronic chest diseases) .

Patient with cerebral palsy.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
Behavioural changes among asthmatic children | 1 year
  evalaution of anaxiety , deppresion and ADHD in asthmatic childern by using psychological tests as ADHD test and IQ test

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Feitosa CA, Santos DN, Barreto do Carmo MB, Santos LM, Teles CA, Rodrigues LC, Barreto ML. Behavior problems and prevalence of asthma symptoms among Brazilian children. J Psychosom Res. 2011 Sep;71(3):160-5. doi: 10.1016/j.jpsychores.2011.02.004. Epub 2011 Mar 21. PMID 21843751
- [Background] Achenbach TM, Ivanova MY, Rescorla LA, Turner LV, Althoff RR. Internalizing/Externalizing Problems: Review and Recommendations for Clinical and Research Applications. J Am Acad Child Adolesc Psychiatry. 2016 Aug;55(8):647-56. doi: 10.1016/j.jaac.2016.05.012. Epub 2016 May 31. PMID 27453078
- [Background] Annett RD, Bender BG, Lapidus J, Duhamel TR, Lincoln A. Predicting children's quality of life in an asthma clinical trial: what do children's reports tell us? J Pediatr. 2001 Dec;139(6):854-61. doi: 10.1067/mpd.2001.119444. PMID 11743513
- [Background] McQuaid EL, Kopel SJ, Nassau JH. Behavioral adjustment in children with asthma: a meta-analysis. J Dev Behav Pediatr. 2001 Dec;22(6):430-9. doi: 10.1097/00004703-200112000-00011. PMID 11773808